CLINICAL TRIAL: NCT02181764
Title: A Phase 1, Multicenter, Open-label, Sequential Dose-escalation, Single-dose Study to Assess the Safety and Tolerability of KRN23 in Subjects With X-linked Hypophosphatemic Rickets/Osteomalacia.
Brief Title: A Study of KRN23 in Subjects With X-linked Hypophosphatemic Rickets/Osteomalacia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kyowa Kirin Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KRN23-001
Record Dates: First submitted 2014-07-02; First posted 2014-07-04 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-02

CONDITIONS: X-linked Hypophosphatemic Rickets/Osteomalacia
Keywords: XLH
MeSH Terms: conditions — Familial Hypophosphatemic Rickets; Osteomalacia | interventions — burosumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- KRN23 (Experimental): Single SC administration on day 1
  Interventions: Drug: KRN23

INTERVENTIONS:
Drug: KRN23 — Single SC administration on day 1: 0.3, 0.6 and 1.0 mg/kg

SUMMARY:
The objective of this study is to assess the safety and tolerability of KRN23 after a single subcutaneous (SC) administration in subjects with X-linked hypophosphatemic rickets/osteomalacia (XLH) in Japan or Korea.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years or older
2. Patients with XLH

Exclusion Criteria:

1. Have an active infection or chronic inflammatory disease
2. Have uncontrolled hypertension
3. Have uncontrolled diabetes mellitus
4. History of known immunodeficiency
5. Use of a pharmacologic vitamin D metabolite or its analogs within 21 days prior to screening and after screening
6. Use of phosphate, calcium preparation, calcimimetics, aluminum hydroxide antacids, thiazide diuretic, acetazolamide, or phosphate, calcium, and/or vitamin D-containing supplements within 10 days prior to screening and after screening
7. Pregnant or lactating females, women who are possibly pregnant or patients who have no intention of utilizing adequate contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Number and types of adverse events | Up to 7 weeks after dosing
  The safety of KRN23 assessed by number and types of adverse events, laboratory tests

SECONDARY OUTCOMES:
Profiles of pharmacokinetics | Pre-dose, 24, 48, 96, 168, 336, 504, 672, 840, 1176 hours post-dose

CONTACTS AND LOCATIONS:
Locations (2):
- Tokyo, Japan
- Seoul, South Korea